CLINICAL TRIAL: NCT03226795
Title: Improving Therapeutic Adherence of Adult Patients With Cystic Fibrosis: Impact of a Co-constructed Program by Patients and Health Caregivers.
Brief Title: Improving Therapeutic Adherence With a Co-constructed Program Involving Both Patients and Health Care Professionals
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 69HCL17_0279
Record Dates: First submitted 2017-07-17; First posted 2017-07-24 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; Therapeutic adherence; Co-constructed intervention; Patient involvement
MeSH Terms: conditions — Cystic Fibrosis; Treatment Adherence and Compliance; Patient Participation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- interventional arm (Experimental)
  Interventions: Other: " Information-Motivation-Behavioral skills " intervention.

INTERVENTIONS:
Other: " Information-Motivation-Behavioral skills " intervention. — * "information" -> Reminders of medication: mobile application
  * "Motivation" -> Coaching by patients: intervention or coaching by an expert patient, animation of a social network of patients
  * "Behavioral skills" -> Accompaniment by professionals: therapeutic education, assessment of membership during medical visits, prioritization of treatments

SUMMARY:
Background Cystic fibrosis is a life-threatening genetic disorder responsible for pulmonary failure and multi-systemic complications involving specific and large medical care burden. To date, no program has shown its effectiveness in improving therapeutic adherence. A new approach to develop a co-constructed program involving patients and professionals may contribute to improve therapeutic adherence.

Objectives The aim of the MUCOBS-Trial project is to create a program to increase therapeutic adherence and to evaluate its efficacy in adult patients with cystic fibrosis in 3 CF centers in France.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Cystic Fibrosis
* Aged 18 or more
* Speaking / understanding French
* Followed in one of the participating centers (CRCM of the Auvergne-Rhône-Alpes region)
* Resident in Auvergne-Rhône-Alpes
* Affiliated to the general health insurance scheme

Exclusion Criteria:

* Transplanted Patients
* Patients who participated in the working group for the co-construction of the intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2021-01-18 (Actual); Primary Completion 2023-04-18 (Estimated); Study Completion 2025-10-18 (Estimated)

PRIMARY OUTCOMES:
Medication Adherence (coverage rate) | 18 months.
  Continuous multiple-interval measures of medication availability (CMA), including:
  * Medications for obstructive airway syndromes
  * Aerosolized bronchial fluidifier
  * Inhaled antibiotics
  * Vitamins
  * Hepatic and biliary therapeutics
  * Pancreatic enzyme replacement therapy
  * Medicinal products for acid disorders
  * Diabetes medications these measurements (coverage rate for each therapeutic class) will be aggregated to evaluate the medication adherence.

SECONDARY OUTCOMES:
Adherence to medications for obstructive airway syndromes | 18 months.
  Continuous multiple-interval measures of medication availability (CMA) for Medications for obstructive airway syndromes
Adherence to physiotherapy | 18 months
  Ratio between the number of acts refunded by the Health Insurance and the theoretical number of acts necessary for compliance with the prescription.
Adherence score evaluated by self-administered questionnaire | 6 and 18 months
  Measured from a self-administered questionnaire, adapted from the Cystic Fibrosis Compliance questionnaire
Cystic Fibrosis Knowledge Scale | 6 and 18 months
  Measured from a self-knowledge questionnaire adapted from the Cystic Fibrosis Knowledge Scale
Quality of life measured by Cystic fibrosis Questionnaire (CFQ-R) | 6 and 18 months
  Measured by Cystic fibrosis Questionnaire (CFQ-R) specific to cystic fibrosis and validated in French
Clinical evolution : Forced expiratory volume in 1 s as a percentage of predicted (%FEV1) | 18 months
  Forced expiratory volume in 1 s as a percentage of predicted (%FEV1) and body mass index (BMI) will be collected during the patient's usual follow-up, on the observational and interventional phases
Clinical evolution : body mass index (BMI) | 18 months
  Body mass index (BMI) will be collected during the patient's usual follow-up, on the observational and interventional phases

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CRCM mixte, Hôpital Estaing, Clermont-Ferrand
  - CRCM Adulte CHU Grenoble Alpes, La Tronche
  - Centre de Ressources et de Compétences de la Mucoviscidose adulte de Lyon - Centre Hospitalier Lyon Sud, Pierre-Bénite